CLINICAL TRIAL: NCT01985997
Title: Postmarketing Safety Study of Q/LAIV in Subjects 2 Through 49 Years of Age
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-VA-MEDI3250-1115
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Observation Safety
Keywords: FluMist, Quadrivalent, Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational post-marketing study conducted in children and adults immunized with Q/LAIV as part of routine clinical practice at Kaiser Permanente Northern California (NCKP) sites.

DETAILED DESCRIPTION:
Children and adults will be immunized with Q/LAIV as part of routine clinical practice at Kaiser Permanente Northern California (NCKP) sites. Using existing data on healthcare utilization, rates of medically attended events (MAEs) of interest will be evaluated in all eligible Q/LAIV recipients who are vaccinated in the Kaiser Permanente (KP) Northern California Health Care Plan during the 2013-2014 influenza season. Enrollment must include a minimum of 10,000 children 2 through 8 years of age; based on previous utilization of FluMist at NCKP, enrollment is expected to include approximately 80,000 children and adults 2 to 49 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. . Age 2 through 49 years at the time of vaccination (or index date for unvaccinated controls)
2. . Membership in the KP Health Care Plan for at least 12 months prior to vaccination/index date
3. . Continuous enrollment in KP Health Care Plan through 6 months following vaccination/index date.

Exclusion Criteria:

NONE

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults 2 to 49 years of age vaccinated with Q/LAIV, TIV or no vaccine at Kaiser Permenente Northern California sites.
Sampling Method: Non-Probability Sample
Enrollment: 95000 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rates of medically attended events: hypersensitivity, seizures/convulsions | From 0-3 days
  Rates of medically attended events from 0 to 3 days: hypersensitivity, seizures/convulsions
Rates of medically attended events: lower respiratory tract infection, wheezing, Guillain-Barré syndrome, Bell's palsy, encephalitis, neuritis, vasculitis, any hospitalization and respiratory hospitalizations | From 1 to 42 days
  Rates of medically attended events from 1 to 42 days: lower respiratory tract infection, wheezing, Guillain-Barré syndrome, Bell's palsy, encephalitis, neuritis, vasculitis, any hospitalization and respiratory hospitalizations
Rates of medically attended events: narcolepsy/cataplexy | From 1 to 180 days
  Rates of medically attended events from 1 to 180 days: narcolepsy/cataplexy

CONTACTS AND LOCATIONS:
Overall Officials: Herve Caspard, MD, Study Director — MedImmune LLC
Locations (1):
- Research Site, Oakland, California, United States

REFERENCES:
- [Derived] Baxter R, Eaton A, Hansen J, Aukes L, Caspard H, Ambrose CS. Safety of quadrivalent live attenuated influenza vaccine in subjects aged 2-49years. Vaccine. 2017 Mar 1;35(9):1254-1258. doi: 10.1016/j.vaccine.2017.01.062. Epub 2017 Feb 2. PMID 28162825
- See also: MA-VA-MEDI3250-1115 Redacted CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1876&filename=MEDI1115%20CSR%20Synopsis%20FINAL%2002Sept2016.pdf